CLINICAL TRIAL: NCT05416021
Title: A Phase I, Open-Label, Randomized, Crossover Trial to Investigate the Relative Bioavailability of the 25 mg Dapivirine Vaginal Ring-004 Inserted Every 30 Days and 100 mg DPV Ring-008 Inserted for 90 Days in Healthy Female Participants
Brief Title: Relative Bioavailability Trial of Dapivirine Ring-004 and Ring-008
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IPM 054
Record Dates: First submitted 2022-04-14; First posted 2022-06-13 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Dapivirine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two treatment sequences (AB or BA). During two consecutive 90-day treatment periods, the participants will receive each of the following treatments according to their assigned treatment sequence. The treatment periods will be separated by a 28-day washout period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 25 mg dapivirine ring (Active Comparator): 25 mg dapivirine vaginal ring (Ring-004) for 90 days (replaced every 30 days) (Treatment A), followed by the 100 mg dapivirine ring (Ring-008) used continuously for 90 days (Treatment B)
  Interventions: Drug: dapivirine
- 100 mg dapivirine ring (Active Comparator): 100 mg dapivirine vaginal ring (Ring-008) used continuously for 90 days (Treatment B), followed by the 25 mg dapivirine ring (Ring-004) for 90 days (replaced every 30 days) (Treatment A)
  Interventions: Drug: dapivirine

INTERVENTIONS:
Drug: dapivirine — dapivirine vaginal ring

SUMMARY:
A Phase I, Open-Label, Randomized, Crossover Trial to Investigate the Relative Bioavailability of the 25 mg Dapivirine Vaginal Ring-004 inserted every 30 days and 100 mg Dapivirine Vaginal Ring-008 inserted for 90 days in Healthy Female Participants

DETAILED DESCRIPTION:
IPM 054 is a Phase I, open-label, randomized, crossover trial to determine the relative bioavailability in plasma and vaginal fluid of two formulations of the dapivirine vaginal ring in HIV-negative women. The trial will compare the dapivirine concentrations achieved in plasma and vaginal fluid over all timepoints for each 90-day use period in a two-period, two-sequence, crossover design.

Participants will be randomized to one of two treatment sequences (AB or BA). During two consecutive 90-day treatment periods, the participants will receive each of the following treatments according to their assigned treatment sequence. The treatment periods will be separated by a 28-day washout period.

Treatment Sequence 1:

• 25 mg dapivirine ring (Ring-004) for 90 days (replaced every 30 days) (Treatment A), followed by the 100 mg dapivirine ring (Ring-008) used continuously for 90 days (Treatment B)

Treatment Sequence 2:

• 100 mg dapivirine ring (Ring-008) used continuously for 90 days (Treatment B), followed by the 25 mg dapivirine ring (Ring-004) for 90 days (replaced every 30 days) (Treatment A)

ELIGIBILITY:
Inclusion Criteria:

1. Assigned female sex at birth per participant report*
2. Age 18 through 45 years (inclusive) at Screening, verified by national identification book/card
3. Able and willing to provide written informed consent to be screened for and enrolled in IPM 054
4. Able and willing to provide adequate locator information for trial retention purposes and be reachable per local standard procedures, eg, by home visit or telephone, or via family or close neighbour contacts (confidentiality to be maintained)
5. Able to complete a diary card
6. Available for all visits and able and willing to comply with all trial procedural requirements
7. Willing to comply with abstinence and other protocol requirements
8. Willing to use male condoms for penile-vaginal intercourse and penile-rectal intercourse for the duration of trial participation
9. Per participant report; using an effective method of contraception for at least 30 days (inclusive) prior to Enrolment, and intending to continue use of an effective method for the duration of trial participation; effective methods include:

   1. hormonal methods (except a contraceptive ring)
   2. intrauterine device (IUD); with no vaginal or gynaecological complaints associated with its use prior to enrolment
   3. sterilisation of participant at least 3 months prior to enrolment Note: Women not at risk of becoming pregnant by virtue of having had a partial hysterectomy or having sex exclusively with cisgender women may be enrolled.
10. In general good health as determined by the Investigator/designee at Screening and Enrolment
11. Human Immunodeficiency Virus (HIV)-negative as determined by an HIV test at the time of screening and enrolment
12. Per participant report at Screening, regular menstrual cycles with at least 21 days between menses
13. Per participant report at Screening and Enrolment, states a willingness to refrain from inserting any non-trial vaginal products or objects into the vagina including, but not limited to tampons, spermicides, female condoms, diaphragms, intravaginal rings, vaginal medications, menstrual cups, cervical caps, douches, lubricants, and sex toys (vibrators, dildos, etc.) for the duration of trial participation
14. Upon pelvic examination (using a speculum) at the time of Enrolment, the cervix and vagina appear normal as determined by the Investigator/Physician
15. Willing to refrain from participation in any other research trial for the duration of this trial

Exclusion Criteria:

* 1) Pregnant at Screening or Enrolment or plans to become pregnant during the trial period* 2) Diagnosed with a urinary tract infection (UTI) or reproductive tract infection (RTI) at Screening or Enrolment based on clinical assessment* 3) Diagnosed with an acute sexually transmitted infection (STI) requiring treatment per current local guidelines at Screening such as gonorrhoea (GC), chlamydia trachomatis (CT), trichomonas, and/or syphilis* 4) Has an abnormal cytology finding at screening or clinically apparent Grade 1 or higher pelvic examination finding (observed by trial staff) at Screening or Enrolment, as per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1, March 2017, and/or Addendum (Female Genital Grading Table for Use in Microbicide Studies [Dated November 2007])* 5) Participant report and/or clinical evidence of any of the following:*

  1. Known adverse reaction to any of the trial products (ever)
  2. Chronic and/or recurrent vaginal candidiasis
  3. Misuse of legal and illegal medication or substances in the 12 months prior to Enrolment
  4. Last pregnancy outcome less than 90 days prior to Enrolment
  5. Gynaecologic or genital procedure (eg, tubal ligation, dilation and curettage, piercing) 45 days or less prior to Enrolment Note: Colposcopy and cervical biopsies for evaluation of an abnormal Pap test as well as IUD insertion/removal are not exclusionary.
  6. Currently breastfeeding or planning to breastfeed during the trial period
  7. Participation in any other research trial involving drugs, medical devices, vaginal products or vaccines, in the 60 days prior to Enrolment 6) Completed use of oral pre-exposure prophylaxis (PrEP) for HIV prevention and/or post-exposure prophylaxis (PEP) for potential HIV exposure within one month prior to screening, and/or anticipated use and/or unwillingness to abstain from PrEP during trial participation 7) Has any Grade 1 or higher laboratory abnormalities at the Screening Visit 8) Participant has a positive test for Hepatitis B surface antigen (HBsAg) or is Hepatitis C virus antibody (HCV-Ab) positive 9) Participant has a positive urine drug test or a positive alcohol breath test.

     10) Has any other condition that, in the opinion of the Investigator, would preclude informed consent, make trial participation unsafe, complicate the interpretation of trial outcome data, or otherwise interfere with achieving the trial objectives including any significant uncontrolled active or chronic medical condition 11) Has plans to relocate away from the trial site area after starting the trial and unable to return for trial visits

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Assigned female sex at birth per participant report*
Enrollment: 124 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
To determine the relative bioavailability of Dapivirine Vaginal Ring-008 compared to Dapivirine Vaginal Ring-004 by comparison of dapivirine plasma pharmacokinetic parameters. | during a 90 day use period
  Dapivirine concentrations in plasma, measured at specified timepoints during each 90-day ring use period.

SECONDARY OUTCOMES:
To further characterize the pharmacokinetic profile of Dapivirine Vaginal Ring-008 compared to Dapivirine Vaginal Ring-004 in vaginal fluid | during each 90 days ring use period
  Dapivirine concentrations in vaginal fluid, measured at specified timepoints during each 90-day ring use period, and for 1 day following ring removal. Vaginal fluid samples will be collected using tear test strips at the location of the cervix.
To evaluate the incidence of Grade 1 or higher genitourinary treatment-emergent adverse events and the incidence of Grade 3 or higher treatment-emergent adverse events of the two dapivirine vaginal ring formulations used continuously for 90 days | during each 90 days ring use period
  Evaluating the incidence of treatment-emergent adverse events with severity grades as defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, and/or Addendum 1 (Female Genital Grading Table for Use in Microbicide Studies [Dated November 2007]).
To assess the effects on vaginal flora when using Dapivirine Vaginal Ring-004 and Dapivirine Vaginal Ring-008 formulations used continuously for 90 days | during each 90 days ring use period
  Assessing the effects by evaluating changes in vaginal pH from baseline and the incidence of bacterial vaginosis, assessed by Nugent scores of ≥ 7, determined from vaginal specimens collected for Gram staining.
To characterize the vaginal microenvironment over the course 90 days of ring use. | during a 90 day use period
  The amount of dapivirine released over three 30-day periods (ie, 90 days) for Ring-004 and over 90 days for Ring-008. Residual dapivirine levels in used rings

CONTACTS AND LOCATIONS:
Overall Officials: Anél Dr Pretorius, MB ChB, Principal Investigator — FARMOVS Pty Ltd, Bloemfontein, South Africa
Locations (1):
- FARMOVS, Bloemfontein, South Africa

IPD SHARING:
Plan to Share IPD: No